CLINICAL TRIAL: NCT05415254
Title: A Randomized Open Label Study to Evaluate Efficacy of Calcitriol Supplementation in COVID-19 Patients With Vitamin D Deficiency
Brief Title: Calcitriol Supplementation in COVID-19 Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2022-0072
Record Dates: First submitted 2022-06-10; First posted 2022-06-13 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Vitamin D Deficiency
MeSH Terms: conditions — COVID-19; Vitamin D Deficiency | interventions — Calcitriol

STUDY DESIGN:
Intervention Model Description: treatment group and control group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): calcitriol 0.25ug daily for 10 days + COVID-19 routine treatment
  Interventions: Drug: Calcitriol
- control group (No Intervention): COVID-19 routine treatment

INTERVENTIONS:
Drug: Calcitriol — Calcitriol supplementation orally
  Other Names: Rocaltrol
  Arms: treatment group

SUMMARY:
This is a randomized, open label study to evaluate the efficacy and safety of calcitriol supplementation in COVID-19 patients with vitamin D deficiency.

DETAILED DESCRIPTION:
This is a randomized, open label study to evaluate the efficacy （clinical and laboratory change）and safety （serum calcium） of calcitriol supplementation in COVID-19 patients with vitamin D deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Hospitalized symptomatic COVID-19 patients;
2. COVID-19 nucleic acid Ct value < 28 (both orf1ab gene Ct value and N gene Ct value < 28);
3. Vitamin D deficiency: 25OHD ≤ 20ng/ml;
4. Age: 18-70 years old;

Exclusion Criteria:

1. Asymptomatic COVID-19 patients ；
2. Hypercalcemia;
3. History of primary hyperparathyroidism;
4. History of triple hyperparathyroidism;
5. Patients who are allergic to calcitriol;
6. Pregnant or lactating women;
7. Patients with severe heart or lung diseases or tumor history;
8. Patients already taking vitamin D or its similar preparations;
9. Participants in other interventional clinical studies (including taking paxlovid);
10. Patients with renal insufficiency (eGFR<60ml/min/1.73m2);
11. Patients considered unsuitable for this study by the investigator；

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2022-06-12 (Estimated); Primary Completion 2022-08-19 (Estimated); Study Completion 2022-09-19 (Estimated)

PRIMARY OUTCOMES:
The cycle threshold (Ct) value of COVID-19 nucleic acid after treatment | The 6th day after treatment
  Nucleic acid test of COVID-19

SECONDARY OUTCOMES:
Clinical symptoms changes | The 6th day after treatment
  fever, cough, sore throat，etc
Laboratory examination changes | The 6th day after treatment
  Complete Blood Count， inflammatory markers ，cytokines

CONTACTS AND LOCATIONS:
Overall Officials: Jing Ma, Dr., Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angelidi AM, Belanger MJ, Lorinsky MK, Karamanis D, Chamorro-Pareja N, Ognibene J, Palaiodimos L, Mantzoros CS. Vitamin D Status Is Associated With In-Hospital Mortality and Mechanical Ventilation: A Cohort of COVID-19 Hospitalized Patients. Mayo Clin Proc. 2021 Apr;96(4):875-886. doi: 10.1016/j.mayocp.2021.01.001. Epub 2021 Jan 9. PMID 33714594
- [Background] Wang Z, Joshi A, Leopold K, Jackson S, Christensen S, Nayfeh T, Mohammed K, Creo A, Tebben P, Kumar S. Association of vitamin D deficiency with COVID-19 infection severity: Systematic review and meta-analysis. Clin Endocrinol (Oxf). 2022 Mar;96(3):281-287. doi: 10.1111/cen.14540. Epub 2021 Jul 12. PMID 34160843
- [Background] Pal R, Banerjee M, Bhadada SK, Shetty AJ, Singh B, Vyas A. Vitamin D supplementation and clinical outcomes in COVID-19: a systematic review and meta-analysis. J Endocrinol Invest. 2022 Jan;45(1):53-68. doi: 10.1007/s40618-021-01614-4. Epub 2021 Jun 24. PMID 34165766
- [Background] Elamir YM, Amir H, Lim S, Rana YP, Lopez CG, Feliciano NV, Omar A, Grist WP, Via MA. A randomized pilot study using calcitriol in hospitalized COVID-19 patients. Bone. 2022 Jan;154:116175. doi: 10.1016/j.bone.2021.116175. Epub 2021 Sep 8. PMID 34508882
- See also: Controlling COVID-19 pandemic through hormone calcitriol — http://wjahr.com/home/article_abstract/633